CLINICAL TRIAL: NCT00573053
Title: Effects of Targeting Lower Arterial Oxygen Saturations on the Development of Control of Breathing in Very Preterm Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Ruben E. Alvaro, Associate Professor of Pediatrics, University of Manitoba, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B2007:157
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-01

CONDITIONS: Development of Control of Breathing
Keywords: hypercapneic response; hyperoxic response; breathing pattern; periodic breathing; sighs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High (Active Comparator): Arterial oxygen saturations in the range of 91-95%
  Interventions: Other: Oxygen saturation range
- Low (Experimental): Arterial oxygen saturations in the range of 85-89%
  Interventions: Other: Oxygen saturation range

INTERVENTIONS:
Other: Oxygen saturation range — Maintain functional oxygen saturation range between 91 and 95%
  Arms: High
Other: Oxygen saturation range — Maintain functional arterial oxygen saturations in the range of 85- 89%
  Arms: Low

SUMMARY:
To determine whether targeting lower arterial oxygen saturations from the day of birth alters the early (first 3 months) postnatal development of the control of ventilation and the hypercapnic and hyperoxic responses in very preterm infants.

DETAILED DESCRIPTION:
To measure the effects of baseline oxygenation in extremely low birth weight preterm infants on:

i) The early (first 5 breaths) and late or steady state (3-5 minutes) ventilatory response to CO2 ii) The immediate (< 1 minute) ventilatory response to hyperoxia iii) The PCO2 apneic threshold iv) The breathing pattern during quiet and REM sleep v) The morphology of periodic breathing cycles vi) The incidence and morphology of sighs

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 23 0/7 - 27 6/7 weeks
* Enrolled in the COT trial at the Health Sciences Centre and the St. Boniface General Hospital in Winnipeg
* Postnatal age between 21 days and 70 days
* Informed written consent obtained from at least one of the parents.

Exclusion Criteria:

* Need for mechanical ventilation, NCPAP or O2
* Sepsis or other known causes of apnea.

Ages: 21 Days to 70 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Effects of targeting lower arterial oxygen saturations on the development of control of breathing in very preterm infants | 3 months

SECONDARY OUTCOMES:
To measure the effects of baseline oxygenation in extremely low birth weight preterm infants on the ventilatory response to CO2 and O2, the PCO2 apneic threshold, and the baseline breathing pattern | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruben E Alvaro, MD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Science Centre, Winnipeg, Manitoba